CLINICAL TRIAL: NCT01080716
Title: Safety, Immunogenicity, and Efficacy Studies of WRSS1, a Live Attenuated Shigella Sonnei Vaccine Candidate, in Healthy Thai Adults
Brief Title: Safety and Efficacy Study of WRSS1, a Shigella Sonnei Vaccine Candidate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Mahidol University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A-15647; 09-0021 (Other: NIH/DMID); 1609 (Other: WRAIR IRB)
Record Dates: First submitted 2009-12-23; First posted 2010-03-04 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Dysentery; Shigella; Diarrhea
MeSH Terms: conditions — Dysentery; Dysentery, Bacillary; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1/Arm 1 of Study: WRSS1 vaccine (Experimental): WRSS1 is a live attenuated S. sonnei vaccine candidate derived from the Mosely strain of S.sonnei
  Interventions: Biological: Part 1/Arm 1 of Study: WRSS1 vaccine
- Part 1/Arm 2 of Study: Placebo vaccine (Placebo Comparator): Placebo
  Interventions: Biological: Part 1/Arm 2 of Study: Placebo vaccine
- Part 2/Arm 1 of Study: S. sonnei 53G (Experimental): 10 volunteers from Study Arm 1/Part 1 (WRSS1 vaccine) plus 4 alternates from Arm 1/Part 1 are given 53G S. sonnei
  Interventions: Biological: Part 2/Arm 1 of Study: S. sonnei 53G
- Part 2/Arm 2 of Study: S sonnei 53G (Active Comparator): 10 subjects (naïve controls) plus 4 alternates are give 53G S sonnei
  Interventions: Biological: Part 2/Arm 2 of Study: S. sonnei 53G

INTERVENTIONS:
Biological: Part 1/Arm 1 of Study: WRSS1 vaccine — Single, oral dose of WRSS1
  Arms: Part 1/Arm 1 of Study: WRSS1 vaccine
Biological: Part 1/Arm 2 of Study: Placebo vaccine — Placebo vaccine
  Arms: Part 1/Arm 2 of Study: Placebo vaccine
Biological: Part 2/Arm 1 of Study: S. sonnei 53G — Subject from Part 1/Arm 1 of Study are given 53G S. sonnei
  Arms: Part 2/Arm 1 of Study: S. sonnei 53G
Biological: Part 2/Arm 2 of Study: S. sonnei 53G — 10 naïve controls are given S. sonnei 53G
  Arms: Part 2/Arm 2 of Study: S sonnei 53G

SUMMARY:
This study is an inpatient trial to determine the safety, immunogenicity and efficacy of the WRSS1 candidate vaccine in healthy Thai adult volunteers.

DETAILED DESCRIPTION:
This study is designed as 2 parts.

* Part 1 is a blinded, placebo-controlled inpatient trial in a total of 20 volunteers (14 vaccinees and 6 controls) to determine the safety and immunogenicity. Volunteers will be vaccinated with a single oral dose of 104 colony forming unit (cfu) of WRSS1 or placebo given with bicarbonate buffer.
* Part 2 will be started approximately 60 days after WRSS1 vaccination. This part is an inpatient phase II efficacy trial involving a challenge with the S.sonnei 53G of 10 vaccinees from the first part and 10 naïve controls.

ELIGIBILITY:
Inclusion Criteria:

1. 20-40 years old; male or female;
2. General good health as determined by a screening evaluation no greater than 30 days before admission;
3. Normal bowel habits (grade 1-2 stools - no more than one to two stools per day with at least one stool per 2 days;
4. Sexually active females willing to use birth control (birth control pills, injection hormonal contraceptive, implant hormonal contraceptive, hormonal patch, IUD, sterilization for effective contraceptive methods, spermicidal products and barrier methods are considered acceptable)during the entire study (starting from study day -30) and for 3 months after completion of the study (approximately a total of 6 months) or sexually inactive females (no sexual contact). Volunteers who take birth control pills will be required to use additional contraceptive methods for the remaining days of the cycle after discharge from the VTC (alteration of gastrointestinal functions from the oral vaccine or challenge strain may lead to unpredictable efficacy of pills);
5. Will be available and willing to continue participation in the second part of the study if he/she has been randomly selected;
6. Pass the Assessment of Understanding of the consent form.

Exclusion Criteria:

1. An acute or chronic medical condition or a clinically significant abnormality on physical exam that, in the opinion of the investigator, would render vaccination or challenge as unsafe;
2. Current use of iron or zinc supplements within the past 7 days; current use of antacids (H2 blockers, omeprazole, OTC agents) or immunosuppressive drug;
3. Unwillingness to follow the study procedures
4. Currently breastfeeding, pregnant (βHCG +) or planning to become pregnant within 3 months after the completion of the study;
5. Allergy to quinolone, sulfa, and penicillin classes of antibiotics;
6. History of any of the following conditions within the past 10 years:

   * Arthritis (two or more episodes of joint pain and swelling),
   * Gastrointestinal disease (diagnosed by a doctor as having irritable bowel disease, Crohn's disease, ulcerative colitis (biopsy confirmed), celiac disease, stomach or intestinal ulcers), or
   * Dyspepsia (digestion or heartburn requiring medication more than once per week);
7. Lifetime previous history of known/suspected Shigella diarrhea (except for volunteers who receive vaccines from Part 1) ;
8. Lifetime history of, or active gallbladder disease;
9. HLA B27 Ag (+); Anti-HIV (+); HBsAg(+); Anti HCV IgG Ab(+); abnormal screening tests judged to be clinically significant as judged by PI or sub-PI (Values are out of the acceptable abnormal range from the table in the protocol) other than mild anemia in females (Hct = 0.33-0.36);
10. Lifetime history of participation in Shigella study (except for volunteers who receive vaccines from Part 1);
11. Concurrent participation in another experimental vaccine or drug study within the past 30 days(except for volunteers who receive vaccines from part1);
12. Serological positive for Shigella sonnei: anti-Shigella sonnei LPS IgG antibody titer in serum >800 (except for volunteers who receive vaccines from Part 1);
13. Receipt of antimicrobial drugs for any reason or acute illness or fever >=38 oC within 7 days before vaccination or challenge;
14. Individuals with household contacts that are immunocompromised;
15. History of major abdominal surgery or laparotomy for any reason in the past 3 years, or abdominal scar of unclear origin;
16. Presence of significant ova or parasite or Shigella bacteria in the stool;
17. Receipt of any of the following (does not include the WRSS1 vaccine):

    * a licensed live, attenuated vaccine within the 30 days of challenge
    * a licensed subunit or killed vaccine within the 14 days of the challenge
    * a blood product, including immunoglobulin, in the 90 days before the challenge

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ladaporn Bodhidatta, MD, Study Director — Department of Enteric Diseases, Armed Forces Research Institute of Medical Sciences; Punnee Pitisuttithum, MBBS, Principal Investigator — Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University; Carl Mason, MD, Study Director — Department of Enteric Diseases, Armed Forces Research Institute of Medical Sciences
Locations (1):
- Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Mahidol University and National Institutes of Health will have access to study data.

REFERENCES:
- [Derived] Pitisuttithum P, Islam D, Chamnanchanunt S, Ruamsap N, Khantapura P, Kaewkungwal J, Kittitrakul C, Luvira V, Dhitavat J, Venkatesan MM, Mason CJ, Bodhidatta L. Clinical Trial of an Oral Live Shigella sonnei Vaccine Candidate, WRSS1, in Thai Adults. Clin Vaccine Immunol. 2016 Jul 5;23(7):564-75. doi: 10.1128/CVI.00665-15. Print 2016 Jul. PMID 27146000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited by contacting people from a list of potential volunteers from previous studies, by friend to friend contact, by internal announcement or by presentation booth in the university, community or blood donor sites. Recruitment and screening was performed by the staff at the Vaccine Trial Center, Mahidol University.
Pre-assignment Details: Part 1 - total of 20 volunteers (14 vaccinees and 6 controls) Part 2 - was started approximately 60 days after WRSS1 vaccination. 10 vaccinees from part 1 and 10 naïve controls
Groups:
- Arm 1: WRSS1 Vaccine: WRSS1 is a live attenuated S. sonnei vaccine candidate derived from the Mosely strain of S. sonnei
- Arm 1: Placebo Vaccine: Placebo comparator
- Arm 2: S. Sonnei 53G: 10 volunteers from Study Arm 1/Part 1 (WRSS1 vaccine) given S. sonnei 53G
- Arm 2: S. Sonnei 53G (Naive Subjects): 10 naïve controls given S. sonnei 53G
Period: Part 1
Arm/Group | Arm 1: WRSS1 Vaccine | Arm 1: Placebo Vaccine | Arm 2: S. Sonnei 53G | Arm 2: S. Sonnei 53G (Naive Subjects)
Started | 14 | 6 | 0 | 0
Completed | 13 | 6 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Arm 1: WRSS1 Vaccine | Arm 1: Placebo Vaccine | Arm 2: S. Sonnei 53G | Arm 2: S. Sonnei 53G (Naive Subjects)
Started | 0 | 0 | 10 | 10
Completed | 0 | 0 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1/Arm 2 of Study: Placebo Vaccine: Placebo comparator
- Part 2/Arm 1 of Study: S. Sonnei 53G: 10 volunteers from Study Arm 1/Part 1 (WRSS1 vaccine) given 53G S. sonnei
- Part 2/Arm 2 of Study: S Sonnei 53G (Controls): 10 subjects (naïve controls) given S. sonnei 53G
- Total: Total of all reporting groups
Arm/Group | Part 1/Arm 1 of Study: WRSS1 Vaccine | Part 1/Arm 2 of Study: Placebo Vaccine | Part 2/Arm 1 of Study: S. Sonnei 53G | Part 2/Arm 2 of Study: S Sonnei 53G (Controls) | Total
Number analyzed (Participants) | 13 | 6 | 10 | 10 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 6 | 10 | 10 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject withdrawn due to diarrhea and mucus in stool prior to vaccination
  Participants
    Female | 8 | 3 | 5 | 2 | 18
    Male | 5 | 3 | 5 | 8 | 21
Region of Enrollment [Number; unit: participants]
  Thailand | 13 | 6 | 10 | 10 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Overview of AEs highlighting all AEs, withdrawals and deaths related to AEs
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1/Arm 1 of Study: WRSS1 Vaccine | Part 1/Arm 2 of Study: Placebo Vaccine | Part 2/Arm 1 of Study: S. Sonnei 53G | Part 2/Arm 2 of Study: S Sonnei 53G (Controls)
Number analyzed (Participants) | 13 | 6 | 10 | 10
Participants
  All Adverse Events | 9 | 5 | 8 | 10
  All Serious Adverse Events | 0 | 0 | 0 | 0
  Withdrawals Due to Adverse Events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Shigella Induced Clinical Disease in Part 2
Description: Study Part 2-Frequency of Shigella induced clinical disease defined as one or more of diarrhea, dysentery or fever in vaccinees and controls following challenge with S. sonnei 53G. Transmissibility of disease will be evaluated by the presence of fecal shedding in control subjects.
Time Frame: 0-5 days
Population: Number of participants in vaccine and controls following the challenge who experienced one or more clinical disease criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2/Arm 1 of Study: S. Sonnei 53G | Part 2/Arm 2 of Study: S Sonnei 53G (Controls)
Number analyzed (Participants) | 10 | 10
Participants
  Diarrhea: Yes | 1 | 1
  Diarrhea: No | 9 | 9
  Dysentery: Yes | 2 | 2
  Dysentery: No | 8 | 8
  Fever: Yes | 1 | 2
  Fever: No | 9 | 8
  Abdominal Pain: Yes | 1 | 2
  Abdominal Pain: No | 9 | 8
  Tenesmus: Yes | 1 | 2
  Tenesmus: No | 9 | 8
  Nausea: Yes | 1 | 1
  Nausea: No | 9 | 9
  Vomiting: Yes | 0 | 1
  Vomiting: No | 10 | 9
  Myalgia: Yes | 2 | 2
  Myalgia: No | 8 | 8
  Joint Pain: Yes | 0 | 0
  Joint Pain: No | 10 | 10
  Dizziness: Yes | 2 | 2
  Dizziness: No | 8 | 8
  Anorexia: Yes | 1 | 1
  Anorexia: No | 9 | 9
  Malaise: Yes | 3 | 2
  Malaise: No | 7 | 8
  Headache: Yes | 2 | 1
  Headache: No | 8 | 9
  Meet Criteria of Clinical Disease: Yes | 3 | 3
  Meet Criteria of Clinical Disease: No | 7 | 7
  Meet Criteria by External Review: Yes | 3 | 6
  Meet Criteria by External Review: No | 7 | 4
  Shedding S.sonnei (Fecal): Yes | 6 | 7
  Shedding S.sonnei (Fecal): No | 4 | 3

3. Secondary Outcome: Count of Subjects With Normal and Abnormal Clinical Laboratory Values During Parts 1 and 2 of Study
Description: Count of subjects in Parts 1 and 2 with normal and abnormal clinical laboratory values after samples taken on days 1, 7, 14, and 28. Abnormal lab values are determined clinically significant by the PI
Time Frame: Days 1, 7, 14, and 28
Population: Count of subjects in Parts 1 and 2 with normal and abnormal clinical laboratory values after samples taken on days 1, 7, 14, and 28. Abnormal lab values are determined clinically significant by the PI. Results were not presented per arm in the FCSR, but were instead presented as parts 1 and 2 of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects From Part 1 of Study: Analysis of abnormal clinical laboratory values in subjects from Part 1 of study
- Subjects From Part 2 of Study: Analysis of abnormal clinical laboratory values in subjects from Part 2 of study
Arm/Group | Subjects From Part 1 of Study | Subjects From Part 2 of Study
Number analyzed (Participants) | 20 | 20
Participants
  Not Clinically Abnormal | 20 | 19
  Clinically Abnormal | 0 | 1

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Part 1/Arm 2: Placebo: Placebo comparator
Arm/Group | Part 1/Arm 1 of Study: WRSS1 Vaccine | Part 1/Arm 2: Placebo | Part 2/Arm 1 of Study: S. Sonnei 53G | Part 2/Arm 2 of Study: S Sonnei 53G (Controls)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/13 | 5/6 | 8/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1/Arm 1 of Study: WRSS1 Vaccine (N=13) | Part 1/Arm 2: Placebo (N=6) | Part 2/Arm 1 of Study: S. Sonnei 53G (N=10) | Part 2/Arm 2 of Study: S Sonnei 53G (Controls) (N=10)
Diarrheic stool (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2) — Mild
Water stool (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 6 (6) — Mild
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) — Mild
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Headache (Nervous system disorders) | 8 (8) | 2 (2) | 4 (4) | 2 (2) — Mild
Tenderness at digit of left foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Moderate
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) — Mild
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5) — Mild
Urticaria (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mild
Insomnia (sleep difficulty) (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Mild
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Moderate
Abrasion wound at peri-anal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Mild
Lower abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Myalgia at back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Mild
Abdominal pain (epigastrium) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Common cold (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) — Mild
Feverish (General disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) — Mild
Pruritus at left thigh (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Abdominal pain (generalized) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Tenesmus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — Mild
Malaise (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) — Mild
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild
Nasal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Myalgia at neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) — Mild
Dysentery (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) — Mild
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Moderate
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) — Mild
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Mild
Chills (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Mild
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Mild
Herpes (lip) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Abdominal pain (whole) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Mild
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
High ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Aphthous (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Tendinitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Increased bowel sound (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild
Perianal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Moderate
Shigellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Severe
Myalgia at right shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No